CLINICAL TRIAL: NCT01199731
Title: A Phase 2b Study to Select a Once Daily Oral Dose of GSK2248761 in HIV-1 Infected Antiretroviral Therapy Experienced Adults With Non-nucleoside Reverse Transcriptase Inhibitor (NNRTI) Resistance
Brief Title: Dose-finding Study of GSK2248761 in Antiretroviral Therapy-experienced Subjects With NNRTI-resistant HIV Infection
Acronym: SONNET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to safety concerns
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113399
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2017-10-12 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: raltegravir; NNRTI; ritonavir; darunavir; HIV; GSK2248761; antiretroviral; HIV Infection; HAART
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — IDX 899; etravirine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK2248761 100mg OAD (Experimental): In combination with darunavir/ritonavir BID and raltegravir BID
  Interventions: Drug: GSK2248761 100 mg once daily
- GSK2248761 200mg OAD (Experimental): In combination with darunavir/ritonavir BID and raltegravir BID
  Interventions: Drug: GSK2248761 200 mg once daily
- Etravirine (Active Comparator): In combination with darunavir/ritonavir BID and raltegravir BID
  Interventions: Drug: Etravirine

INTERVENTIONS:
Drug: GSK2248761 100 mg once daily — 1 100mg capsule OAD plus matching placebo
  Arms: GSK2248761 100mg OAD
Drug: GSK2248761 200 mg once daily — 2 100mg capsules OAD
  Arms: GSK2248761 200mg OAD
Drug: Etravirine — 2 100mg tablets twice daily
  Arms: Etravirine

SUMMARY:
This 48 week, phase 2b study in 150 HIV-1 infected antiretroviral therapy experienced adult subjects consists of a dose-ranging evaluation of GSK2248761 at blinded doses of 100 mg and 200 mg once daily with a control arm of open-label etravirine (ETV) 200 mg twice daily. The background ART for all three arms will be darunavir/ritonavir (DRV/r) 600 mg/100 mg twice daily plus raltegravir (RAL) 400 mg twice daily. Antiviral activity, safety, PK, and development of viral resistance will be evaluated.

DETAILED DESCRIPTION:
Study SGN113399 is a Phase 2b randomized, partially-blinded, multicenter, parallel-group, dose-ranging study to be conducted in HIV-1 infected ART-experienced adults with documented NNRTI resistance.

A minimum of 150 subjects will be randomized 1:1:1 to one of two GSK2248761 doses or a control regimen containing ETV (50 subjects per group); all subjects will also receive darunavir/ritonavir and raltegravir. The trial will be partially blinded, i.e. subjects receiving GSK2248761 and the investigators will be blinded to the dose they receive. Subjects will not be blinded to whether they receive GSK2248761 or ETV.

Randomization will be stratified by:

* HIV-1 VL at screening, <50,000 copies/mL or >/50,000 copies/mL, and
* Darunavir susceptibility (screening phenotype fold change <7 or >/7 to 20)

Background ART will be administered open-label.

The primary endpoint analysis will take place after all subjects have completed Week 16. An optimal dose of GSK2248761 will be determined by the Week 16 analysis; this dose selection will be confirmed using an analysis from all subjects following completion of Week 24. If there is a clear efficacy, safety or tolerability advantage driving dose selection for GSK2248761, then all subjects receiving the non-selected dose of GSK2248761 will be switched to the selected dose following dose confirmation, after all subjects have completed Week 24. If no differentiation of dose can be made based on objective measures of efficacy, safety or tolerability, then both doses will be continued through Week 48.

After Week 48, all subjects will be expected to obtain local access to all commercially available ART.

No regimen switches of either background ART (DRV/r and RAL) or test agent or control (GSK2248761 and ETV) are allowed during the 48 week period of the study.

Study Endpoints/Assessments Subjects will have assessments performed which will include baseline demographics, disease characteristics, pharmacogenetics (PGx) and safety (laboratory and clinical evaluations). On study safety, efficacy, virologic, immunologic, and PK evaluations will also be conducted.

The primary endpoint will be the proportion of subjects with HIV-1 RNA <50copies/mL at Week 16. Dose selection will be based primarily on antiviral activity and tolerability in conjunction with immunologic, safety, virologic resistance and PK measures. Data from the Week 24 analysis will be used to confirm dose selection.

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adults greater than or equal to 18 years of age. Females are eligible to enter and participate in the study if she is (1) non-childbearing potential, (2) child bearing potential with negative pregnancy test at screening and Day 1 and agrees to use protocol-specified methods of birth control while on study.
* HIV-1 infection with a screening plasma HIV-1 RNA greater than or equal to 400copies/mL
* Previously received or current treatment with antiretroviral therapy (HAART) for HIV-1 infection (patient may be off ART at time of screening)
* HIV-1 harboring NNRTI resistance by screening genotype (defined as the presence of at least 1 NNRTI resistance-associated mutations)

Exclusion Criteria:

* Any pre-existing physical or mental condition (including substance abuse disorder) which, in the opinion of the Investigator, may interfere with the subject's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the subject
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the drug or render the subject unable to take oral medication
* Women who are currently breastfeeding
* Any evidence of an active Centers for Disease and Prevention Control (CDC) Category C disease [CDC, 1993], except cutaneous Kaposi's sarcoma not requiring systemic therapy
* History of ongoing or clinically relevant hepatitis within the previous 6 months, including chronic hepatitis B virus (HBV) infection (HBsAg positive). Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded, however Investigators must carefully assess if therapy specific for HCV infection is required; subjects who are anticipated to require such therapy during the randomized portion of the study must be excluded
* History of liver cirrhosis with or without hepatitis viral co-infection
* Ongoing or clinically relevant pancreatitis
* History of the following cardiac diseases: myocardial infarction, congestive heart failure, documented hypertrophic cardiomyopathy, sustained ventricular tachycardia
* Personal or known family history of prolonged QT syndrome
* History or presence of allergy or intolerance to the study drugs or their components, or a history of drug or other allergy that, in the opinion of the Principal Investigator, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled
* HIV-1 genotype results with any of the following will be excluded: (1)Any screening genotype with virus showing a Y181 mutation in combination with any other NNRTI resistance-associated mutations, (2) Any screening genotype with virus showing a Y181I or Y188L alone or in combination with any other NNRTI resistance-associated mutations
* HIV-1 phenotype results with any of the following will be excluded: (1) Any screening phenotype with virus showing etravirine fold change >10, (2) Any screening phenotype with virus showing darunavir fold change > 20, (3) Any screening phenotype with virus showing raltegravir fold change >1.5
* Any acute laboratory abnormality at screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study of an investigational compound. Any verified Grade 4 laboratory abnormality at screening would exclude a subject from study participation unless the Investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the medical monitor
* Any of the following laboratory values at screening: (1) Creatinine clearance <50 mL/min via Cockroft-Gault method, (2) Alanine aminotransferase (ALT) greater than or equal to 5 times ULN. Subjects with ALT >2xULN but <5xULN may participate in the study, if in the opinion of the Investigator and GSK medical monitor the lab abnormality will not interfere with the study procedures or compromise subject safety, (3) Alanine aminotransferase (ALT) greater than or equal to 3xULN and bilirubin greater than or equal to 1.5xULN (with >35% direct bilirubin
* Any clinically significant finding on screening electrocardiograph (ECG), specifically (a single repeat is allowed to determine eligibility): (1) Heart rate <45 and >100bpm (males), <50 and >100bpm (females); Note: A heart rate from 100 to 110 BPM can be rechecked within 30 minutes to verify eligibility, (2) QRS duration >120msec, (3) QTc interval >450msec, (4) Non-sustained (greater than or equal to 3 consecutive beats) or sustained ventricular tachycardia, (5) Sinus pauses >2.5 seconds, (6) 2nd degree (Type II) or higher AV (Atrioventricular) block, (7) Evidence of WPW (Wolff-Parkinson-White) syndrome (ventricular preexcitation), (8) Pathologic Q waves (defined as Q wave >40msec OR depth >0.4 mV, (9) Any other abnormality which in the opinion of the investigator would interfere with the safety of the subject
* Treatment with any of the following agents within 28 days prior to screening, or has an anticipated need for these agents during the study: (1) radiation therapy or cytotoxic chemotherapeutic agents, (2) immunomodulators (such as systemic corticosteroids, interleukins, or interferons); Note: Subjects using short-term (<7 day) steroid tapers and inhaled corticosteroids are eligible for enrollment, (3) Any non-protocol-specified agent with documented activity against HIV-1 in vitro
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days prior to screening
* Receipt of an experimental drug and/or vaccine within 28 days or 5 half-lives, or twice the duration of the biological effect of the experimental drug or vaccine, whichever is longer, prior to screening
* Immunization within 28 days prior to first dose of IP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10-05 (Actual); Primary Completion 2011-07-19 (Actual); Study Completion 2011-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (36):
- United States (28):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Longview, Texas
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Liège
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Italy (2):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Monza, Lombardy
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Constanța

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 investigational sites enrolled participants in this multicenter study: 1 center in Romania and 16 in the United States. The study was initiated on 04 October 2010 and was terminated on 01 April 2011 with last participant visit on 19 July 2011.
Pre-assignment Details: Enrollment in this study was terminated prematurely due to a safety finding (convulsions) in 5/20 participants who received GSK2248761. At time of enrollment termination, 30/150 planned participants were enrolled.
Groups:
- GSK2248761 100 Milligram (mg): Participants received GSK2248761 1 x 100 mg capsule once daily orally, 1 x Placebo to match GSK2248761 capsule once daily orally, Darunavir (DRV) 1 x 600 mg tablet twice daily with food orally, Ritonavir (RTV) 1 x 100 mg tablet twice daily orally and Raltegravir(RAL) 1 x 400 mg tablet twice daily orally up to 48 weeks.
- GSK2248761 200 mg: Participants received GSK2248761 2 x 100 mg capsule once daily orally, DRV 1 x 600 mg tablet twice daily with food orally, RTV 1 x 100 mg tablet twice daily orally and RAL 1 x 400 mg tablet twice daily orally up to 48 weeks.
- Etravirine (ETV): Participants received ETV 2 x 100 mg tablet once daily orally, DRV 1 x 600 mg tablet twice daily with food orally, RTV 1 x 100 mg tablet twice daily orally and RAL 1 x 400 mg tablet twice daily orally up to 48 weeks.
Period: Overall Study
Arm/Group | GSK2248761 100 Milligram (mg) | GSK2248761 200 mg | Etravirine (ETV)
Started | 9 | 11 | 10
Completed | 0 | 0 | 0
Not Completed | 9 | 11 | 10
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Study closed/terminated | 7 | 9 | 7
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK2248761 100 mg: Participants received GSK2248761 1 x 100 mg capsule once daily orally, 1 x Placebo to match GSK2248761 capsule once daily orally, DRV 1 x 600 mg tablet twice daily with food orally, RTV 1 x 100 mg tablet twice daily orally and RAL 1 x 400 mg tablet twice daily orally up to 48 weeks.
- ETV 200 mg: Participants received ETV 2 x 100 mg tablet once daily orally, DRV 1 x 600 mg tablet twice daily with food orally, RTV 1 x 100 mg tablet twice daily orally and RAL 1 x 400 mg tablet twice daily orally up to 48 weeks.
- Total: Total of all reporting groups
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg | ETV 200 mg | Total
Number analyzed (Participants) | 9 | 11 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (9.11) | 42.4 (11.60) | 43.2 (8.75) | 43.6 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 9
  Male | 7 | 9 | 5 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 6 | 14
  White | 5 | 5 | 4 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) <50 Copies Per Milliliter (/mL) at Week 16
Description: Plasma for quantitative HIV-1 RNA was collected. The percentage of participants with HIV-1 RNA <50 copies/mL at Week 16 has been presented. A 2 ml plasma was assayed with the real-time NucliSens EasyQ HIV-1 assay (bioMerieux) capable of quantifying as low as 2.5 c/mL by using three modifications to the standard assay: 15 microliters (µl) of extracted eluate, 20 µl of primer, and 5 µl of 2X enzyme in place of standard kit volumes. The validated assay incorporated molecular beacons for detection.
Time Frame: At Week 16
Population: Intent-to-Treat-Exposed (ITT-E) consisted of all randomized participants who received at least one dose of investigational product (IP). Only those participants with data available at the indicated time point were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg | ETV 200 mg
Number analyzed (Participants) | 0 | 0 | 3
Percentage of participants |  |  | 33

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to follow-up i.e. 2-4 weeks after the last study visit (due to early termination the last visit was on 19 July 2011)
Population: Safety population consisted of all randomized participants who were exposed to IPs with the exception of any participant with documented evidence of not having consumed any amount of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg | ETV 200 mg
Number analyzed (Participants) | 9 | 11 | 10
Participants
  Any AE | 7 | 9 | 6
  Any SAE | 1 | 4 | 0

3. Secondary Outcome: Number of Participants With Abnormal Clinical Chemistry Laboratory Data With Grade 3 or 4 Treatment-Emergent (TE) Toxicities
Description: A toxicity was considered to be TE if it was greater than the Baseline grade, and if it had developed or increased post-Baseline in intensity (and prior to the last dose of IP). Division of acquired immunodeficiency syndrome (AIDS) toxicity scale for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0 was used for grading i.e. Grade 3=severe and Grade 4=potentially life threatening. Categories with values have been presented. No toxicity-related dose reductions of IP was allowed. IP and background antiretroviral therapy (ART) was restarted as soon as medically appropriate; in general, this was no longer than 14] days after discontinuation (unless Grade 3 or 4 toxicities persisted).
Time Frame: Up to follow-up i.e. 2-4 weeks after the last study visit (due to early termination the last visit was on 19 July 2011)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg | ETV 200 mg
Number analyzed (Participants) | 9 | 11 | 10
Participants
  Grade 3: Glucose | 1 | 0 | 0
  Grade 3: Hyperglycaemia | 1 | 0 | 0

4. Secondary Outcome: Number of Participants With Abnormal Hematology Laboratory Data With Grade 3 or 4 TE Toxicities
Description: A toxicity was considered to be TE if it was greater than the Baseline grade, and if it had developed or increased post-Baseline in intensity (and prior to the last dose of IP). The hematology parameters included hemoglobin, total neutrophils, and white blood cells (WBC) count. Categories with values has been presented. Grade 3=severe and Grade 4=potentially life threatening. No toxicity-related dose reductions of IP was allowed. IP and background ART was restarted as soon as medically appropriate; in general, this was no longer than 14] days after discontinuation (unless Grade 3 or 4 toxicities persisted).
Time Frame: Up to follow-up i.e. 2-4 weeks after the last study visit (due to early termination the last visit was on 19 July 2011)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg | ETV 200 mg
Number analyzed (Participants) | 9 | 11 | 10
Participants
  Grade 3: Total Neutrophils | 1 | 1 | 0
  Grade 3: WBC | 0 | 1 | 0

5. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA Prior to Switch of GSK2248761
Description: A switch was defined as any ART substitution or addition in the participant's ART regimen. Any ART switch permitted per protocol that was determined necessary and documented prior to the first on-treatment visit where HIV-1 RNA was assessed could occur without penalty. However, any participants with an ART switch not permitted per protocol or ART switch permitted per protocol with a viral load >=50 copies/mL at the time of the decision to switch was made was counted as a non-responder from that point onward for all assessment windows without a viral load measurement collected prior to the switch. Change from Baseline was calculated as (observed value - Baseline value). Baseline was Day 1. The unit is log10 copies per milliliter (log10 copies/mL).
Time Frame: Baseline (Day 1) and Week 2, 4, 8, 12 and 16
Population: ITT-E population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg | ETV 200 mg
Number analyzed (Participants) | 9 | 11 | 10
Log10 copies/mL
  Week 2: number analyzed (Participants) | 8 | 10 | 9
  Week 2 | -1.845 (0.6029) | -2.075 (0.7070) | -1.730 (1.0923)
  Week 4: number analyzed (Participants) | 4 | 6 | 9
  Week 4 | -1.985 (0.6818) | -2.621 (0.5614) | -2.064 (1.2401)
  Week 8: number analyzed (Participants) | 5 | 4 | 9
  Week 8 | -2.332 (1.1915) | -3.030 (0.1170) | -1.850 (1.0895)
  Week 12: number analyzed (Participants) | 3 | 1 | 7
  Week 12 | -1.997 (0.8918) | -3.085 (NA) — Not calculable for single participant | -1.678 (1.7096)
  Week 16: number analyzed (Participants) | 0 | 0 | 3
  Week 16 |  |  | -0.820 (1.6424)

6. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA After Switch of GSK2248761
Description: A switch was defined as any ART substitution or addition in the participant's ART regimen. Any ART switch permitted per protocol that was determined necessary and documented prior to the first on-treatment visit where HIV-1 RNA was assessed could occur without penalty. However, any participants with an ART switch not permitted per protocol or ART switch permitted per protocol with a viral load >=50 copies/mL at the time of the decision to switch was made was counted as a non-responder from that point onward for all assessment windows without a viral load measurement collected prior to the switch. Change from Baseline was calculated as (observed value - Baseline value ). Baseline was Day 1.
Time Frame: Baseline (Day 1) and post switch Week 1, 2, 4, withdrawal and follow-up Week 4, 8, 12
Population: ITT-E. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg
Number analyzed (Participants) | 9 | 11
log10 copies/mL
  Week 1 post switch: number analyzed (Participants) | 6 | 8
  Week 1 post switch | -2.080 (1.2175) | -2.197 (1.0203)
  Week 2 post switch: number analyzed (Participants) | 6 | 7
  Week 2 post switch | -2.376 (1.1765) | -2.229 (1.2522)
  Week 4 post switch: number analyzed (Participants) | 2 | 5
  Week 4 post switch | -1.617 (0.8490) | -2.545 (0.6035)
  Withdrawal: number analyzed (Participants) | 7 | 11
  Withdrawal | -2.070 (1.4825) | -1.978 (1.5884)
  4 Week follow-up: number analyzed (Participants) | 9 | 10
  4 Week follow-up | -2.123 (1.2717) | -1.999 (1.2019)
  8 Week follow-up: number analyzed (Participants) | 8 | 9
  8 Week follow-up | -2.101 (1.3686) | -1.251 (1.3476)
  12 Week follow-up: number analyzed (Participants) | 1 | 3
  12 Week follow-up | 0.278 (NA) — Not calculable for 1 participant | -2.272 (0.7077)

7. Secondary Outcome: Number of Participants Who Experienced Disease Progression (HIV-associated Conditions, AIDS and Death)
Description: Clinical DP was defined as progression from Baseline HIV disease status:Category A at Baseline to Centers for Disease Control and Prevention(CDC) category B event, category A at Baseline to CDC category C event, category B at Baseline to CDC category C event, category C at Baseline to new CDC category C event or category A, B or C at Baseline to death. Category A consisted of one or more of the conditions like asymptomatic HIV infection, persistent generalized lymphadenopathy and acute (primary) HIV infection with accompanying illness in an adolescent or adult(>13 years) with documented HIV infection. Category B consisted like Bacillary angiomatosis, Candidiasis, oropharyngeal (thrush), Candidiasis, vulvovaginal; persistent, frequent, oral, Herpes zoster etc. Category C included clinical conditions listed like Candidiasis of bronchi, trachea, or lungs, Candidiasis, esophageal, Cervical cancer, Coccidioidomycosis, disseminated or extrapulmonary etc in AIDS surveillance case definition.
Time Frame: Up to follow-up i.e. 2-4 weeks after the last study visit (due to early termination the last visit was on 19 July 2011)
Population: ITT-E population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg | ETV 200 mg
Number analyzed (Participants) | 9 | 11 | 10
Participants
  Disease progression | 0 | 0 | 0
  Death | 0 | 0 | 0

8. Secondary Outcome: Absolute Values of CD4+ Cell Counts After Switch of GSK2248761
Description: CD4 is a receptor for the HIV virus. Most of the damage to an AIDS participant's immune system was done by the virus' destruction of CD4+ lymphocytes. Absolute values of CD4+ cell counts after Switch of GSK2248761 has been presented.
Time Frame: Baseline (Day 1) and post switch Week 1, 2, 4, withdrawal and Follow-up Week 4, 8, 12
Population: ITT-E. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter (cells/mm^3)
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg
Number analyzed (Participants) | 9 | 11
Cells per cubic millimeter (cells/mm^3)
  Baseline | 229.2 (131.99) | 162.5 (108.16)
  Baseline switch: number analyzed (Participants) | 4 | 6
  Baseline switch | 311.0 (95.11) | 164.3 (107.79)
  Week 1 post switch: number analyzed (Participants) | 6 | 7
  Week 1 post switch | 253.0 (122.25) | 189.9 (132.13)
  Week 2 post switch: number analyzed (Participants) | 6 | 8
  Week 2 post switch | 263.7 (112.85) | 179.0 (101.59)
  Week 4 post switch: number analyzed (Participants) | 2 | 5
  Week 4 post switch | 471.5 (64.35) | 199.6 (48.72)
  Withdrawal: number analyzed (Participants) | 7 | 11
  Withdrawal | 254.6 (137.11) | 188.5 (95.30)
  Week 4 follow-up: number analyzed (Participants) | 9 | 10
  Week 4 follow-up | 289.0 (154.44) | 237.9 (110.27)
  Week 8 follow-up: number analyzed (Participants) | 8 | 10
  Week 8 follow-up | 277.5 (139.41) | 207.2 (117.79)
  Week 12 follow-up: number analyzed (Participants) | 0 | 3
  Week 12 follow-up |  | 329.3 (159.20)

9. Secondary Outcome: Change From Baseline in CD4+ Cell Counts Prior to Switch of GSK2248761
Description: CD4 is a receptor for the HIV virus. Most of the damage to an AIDS patient's immune system is done by the virus' destruction of CD4+ lymphocytes. Change from Baseline was calculated as (observed value - Baseline value). Baseline was Day 1 value.
Time Frame: Baseline (Day 1) and Week 2, 4, 8, 12 and 16
Population: ITT-E. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg | ETV 200 mg
Number analyzed (Participants) | 9 | 11 | 10
Cells/mm^3
  Week 2: number analyzed (Participants) | 8 | 10 | 9
  Week 2 | 43.0 (65.74) | 21.2 (58.05) | 62.2 (81.88)
  Week 4: number analyzed (Participants) | 4 | 6 | 9
  Week 4 | 122.8 (133.34) | 60.7 (79.66) | 81.4 (96.88)
  Week 8: number analyzed (Participants) | 5 | 4 | 9
  Week 8 | 76.4 (111.61) | 57.3 (54.29) | 71.0 (61.19)
  Week 12: number analyzed (Participants) | 2 | 1 | 6
  Week 12 | 41.0 (21.21) | 30.0 (NA) — Not calculable for 1 participant | 61.5 (91.53)
  Week 16: number analyzed (Participants) | 0 | 0 | 3
  Week 16 |  |  | -7.0 (2.00)

10. Secondary Outcome: Change From Baseline in CD4+ Cell Counts After Switch of GSK2248761
Description: as for outcome 9
Time Frame: Baseline (Day 1) and post switch Week 1, 2, 4, withdrawal and Follow-up Week 4, 8, 12
Population: ITT-E. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg
Number analyzed (Participants) | 9 | 11
Cells/mm^3
  Week 1 post switch: number analyzed (Participants) | 6 | 7
  Week 1 post switch | 48.2 (61.10) | 7.4 (54.99)
  Week 2 post switch: number analyzed (Participants) | 6 | 8
  Week 2 post switch | 58.8 (48.55) | 4.3 (42.28)
  Week 4 post switch: number analyzed (Participants) | 2 | 5
  Week 4 post switch | 74.0 (62.23) | 16.6 (61.59)
  Withdrawal: number analyzed (Participants) | 7 | 11
  Withdrawal | 44.1 (74.26) | 26.0 (71.00)
  4 Week follow-up: number analyzed (Participants) | 9 | 10
  4 Week follow-up | 59.8 (56.62) | 72.0 (102.38)
  8 Week follow-up: number analyzed (Participants) | 8 | 10
  8 Week follow-up | 66.3 (54.09) | 32.3 (34.16)
  12 Week follow-up: number analyzed (Participants) | 0 | 3
  12 Week follow-up |  | 113.7 (63.61)

11. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to AEs
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Time Frame: Up to follow-up i.e. 2-4 weeks after the last study visit (due to early termination the last visit was on 19 July 2011)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg | ETV 200 mg
Number analyzed (Participants) | 9 | 11 | 10
Participants | 0 | 2 | 0

12. Secondary Outcome: Number of Participants With Electrocardiograph (ECG) With Values of Potential Critical Concern (PCI)
Description: Number of participants with ECG of PCI above 480 has been presented. ECG was be performed twice on Day 1 at least 5 minutes apart and following 5 minutes of rest in a semi supine position at ∼1 hour prior to first dose. ECG evaluations at other visits was obtained after dosing, preferably at 2 hours post dosing. An ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and corrected QT (QTc) intervals was used.
Time Frame: Up to follow-up i.e. 2-4 weeks after the last study visit (due to early termination the last visit was on 19 July 2011)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg | ETV 200 mg
Number analyzed (Participants) | 9 | 11 | 10
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to follow-up i.e. 2-4 weeks after the last study visit (due to early termination the last visit was on 19 July 2011)
Description: Safety population was used for the analysis.
Arm/Group | GSK2248761 100 mg | GSK2248761 200 mg | ETV 200 mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/9 | 4/11 | 0/10
Other Adverse Events (participants affected / at risk) | 8/9 | 9/11 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2248761 100 mg (N=9) | GSK2248761 200 mg (N=11) | ETV 200 mg (N=10)
Convulsion (Nervous system disorders) | 0 | 4 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2248761 100 mg (N=9) | GSK2248761 200 mg (N=11) | ETV 200 mg (N=10)
Sinusitis (Infections and infestations) | 3 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Body tinea (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Parkinsonism (Nervous system disorders) | 1 | 0 | 0
Petit mal epilepsy (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Eosinophilic pustular folliculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Enrollment in this study was terminated prematurely on 01 April 2011 due to a safety finding (convulsion) in 5/20 participants receiving GSK2248761.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.